CLINICAL TRIAL: NCT01736215
Title: Prediction of Response to Erythropoietin Treatment in Cancer Related Anemia Patients Receiving Chemotherapy
Brief Title: An Observational Study to Predict the Response of Erythropoietin Treatment in Participants With Cancer Related Anemia Receiving Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: This study was terminated regarding to slow enrollment.
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: CR016558; EPOCAN4028
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Anemia - Cancer Related
Keywords: Anemia - cancer related; Eprex (Erythropoietin alfa)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for hematological analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with cancer related anemia: Participants with cancer related anemia receiving chemotherapy will be observed for response to erythropoietin treatment.
  Interventions: Drug: Erythropoietin: Observational study

INTERVENTIONS:
Drug: Erythropoietin: Observational study — This is an observational study. Participants receiving erythropoietin (dosage and regimen will comply with Thai Food and Drug Administration approval package insert) will be observed.

SUMMARY:
The purpose of this observational study is to evaluate the predictors of response to erythropoietin (hormone secreted by kidney that helps in formation of red blood cells in bone marrow) treatment in participants with cancer (abnormal tissue that grows and spreads in the body until it kills) related anemia (decreased number of red blood cells), receiving chemotherapy (treatment of cancer using drugs).

DETAILED DESCRIPTION:
This is an observational, prospective (study following participants forward in time), multi-center (study conducted in more than 1 center) study to identify the predictive factors that will effectively predict the response to erythropoietin treatment in cancer related anemia participants receiving chemotherapy. The entire duration of study will be approximately 1 year. Participants will primarily be evaluated for achieving at least 1 gram per deciliter (g per dl) rise in hemoglobin (substance that carries oxygen and gives blood its red color) level after receiving erythropoietin treatment based on National Comprehensive Cancer Institute (NCCN) V3.2009 practice guideline criteria. Response to erythropoietin treatment will also be predicted using other independent hematological (related to blood) factors like C-reactive protein (CRP - is an acute serum protein released from liver). It is associated with low hemoglobin [substance that carries oxygen and gives blood its red color] or erythropoietin [hormone secreted by kidney that helps in formation of red blood cells in bone marrow] resistance), erythropoietin (EPO), hemoglobin, hematocrit (amount of red blood cells in blood), reticulocyte (immature red blood cells) count, ferritin (a protein that stores iron and allows the body to use iron), serum iron (iron is in the blood which is bound to transferrin) and transferring iron binding capacity (TIBC), level. Number of blood transfusions and participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-hematologic malignancy (cancer or other progressively enlarging and spreading tumor, usually fatal if not successfully treated)
* Participants with life expectancy of at least 6 months based on the Investigator's clinical judgment
* Participants receiving chemotherapy
* Participants having indication and planning to receiving erythropoietin (dosage and regimen should comply with Thai FDA approval package insert)
* Participants who have given consent form

Exclusion Criteria:

* Participants with anemia due to other factors (i.e., iron, B12 or folate deficiencies, hemolysis [breakdown in red blood cells], gastrointestinal bleeding, or any active bleeding)
* Participants with previous history of erythropoietin treatment
* Participants who have received blood transfusion within 1 month before starting erythropoietin therapy
* Pregnant or breast-feeding female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant with cancer related anemia receiving chemotherapy will be observed for response to erythropoietin treatment.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (3):
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Cancer Related Anemia: Participants with cancer related anemia receiving erythropoietin (dosage and regimen were complied with Thai food and drug administration approval package insert) were observed for response to erythropoietin treatment.
Period: Overall Study
Arm/Group | Participants With Cancer Related Anemia
Started | 33
Treated | 25
Completed | 19
Not Completed | 14
Not completed — Early termination of erythropoietin use | 1
Not completed — Adverse Event | 4
Not completed — Progressive disease stop chemotherapy | 1
Not completed — Insufficient data to perform analysis | 8

BASELINE CHARACTERISTICS:
Population: Number of participants analyzed for this baseline characteristic included all the participants who received erythropoietin treatment and had sufficient data to perform statistical evaluation.
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.20 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Erythropoietin Treatment
Description: Responders of erythropoietin treatment were defined as participants who achieved at least 1 gram per deciliter (g per dl) rise from Baseline in hemoglobin level during within 4-8 weeks or participants who achieved 12 g per dl hemoglobin level at anytime during the study evaluation period (about 8 weeks of follow-up, hemoglobin level reached to 12 g per dl or participants who received blood transfusion at any time of study period) based on National Comprehensive Cancer Institute (NCCN) V3.2009 practice guideline criteria.
Time Frame: 8 weeks
Population: Participants who received erythropoietin treatment and had the data available at least on Baseline and at the end of study evaluation period.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 19
Percentage of participants | 52.63

2. Secondary Outcome: Number of Participants With Serum Erythropoietin (EPO) Level (EPO Less Than or Equal to 45.2 or EPO Greater Than 45.3)
Description: EPO is a hormone secreted by kidney that helps in formation of red blood cells in bone marrow. Number of participants with EPO level less than or equal to 45.2 or greater than 45.3 were observed.
Time Frame: Baseline
Population: Participants who received erythropoietin treatment and who had sufficient data to perform statistical evaluation were analyzed.
Measure: Number; unit: Participants
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 25
Participants
  EPO level less than or equal to 45.2 | 12 (59.05)
  EPO level greater than 45.3 | 13
Statistical Analysis 1: Comparison: Participants With Cancer Related Anemia; Test type: Superiority or Other; p = 0.266, Regression, Logistic — The binary logistic regression analysis was performed using a crude model between predictor variable endogenous EPO (EPO less than or equal to 45.2 and EPO greater than 45.3); Odds Ratio (OR) = 0.343, 95% CI 2-sided [0.052 to 2.261]

3. Secondary Outcome: Number of Participants With C-Reactive Protein (CRP) Level Less Than or Equal to 10.3 or Greater Than 10.4
Description: CRP is a acute serum protein released from liver. It is associated with low hemoglobin or erythropoeitin resistance. Number of participants with CRP level less than or equal to 10.3 or greater than 10.4 were observed.
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 25
Participants
  CRP less than or equal to 10.3 | 13 (27.22)
  CRP greater than 10.4 | 12
Statistical Analysis 1: Comparison: Participants With Cancer Related Anemia; Test type: Superiority or Other; p = 0.05, Regression, Logistic — The binary logistic regression analysis was performed using a crude model between predictor variable CRP (CRP less than or equal to 10.3 and CRP greater than 10.4); Odds Ratio (OR) = 0.125, 95% CI 2-sided [0.016 to 0.999]

4. Secondary Outcome: Serum Hemoglobin Level
Description: Hemoglobin is defined as a substance that carries oxygen and gives blood its red color.
Time Frame: Baseline, Week 1, Week 2, Week 4 and Week 8
Population: Participants who received erythropoietin treatment and had the data available at least on Baseline and at all measurable time points of study evaluation period. Here, 'n' signifies participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Gram per deciliter (g per dl)
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 19
Gram per deciliter (g per dl)
  Baseline (n=19) | 9.96 (0.93)
  Week 1 (n=18) | 9.94 (0.94)
  Week 2 (n=18) | 10.00 (1.06)
  Week 4 (n=18) | 10.64 (1.59)
  Week 8 (n=7) | 10.43 (1.49)

5. Secondary Outcome: Serum Hematocrit Level
Description: Hematocrit is the amount of red blood cells in the blood.
Time Frame: Baseline, Week 1, Week 2, Week 4 and Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 19
Percentage of red blood cells
  Baseline (n=19) | 30.75 (3.34)
  Week 1 (n=18) | 30.59 (2.93)
  Week 2 (n=18) | 30.76 (3.17)
  Week 4 (n=18) | 33.19 (5.41)
  Week 8 (n=7) | 33.01 (5.09)

6. Secondary Outcome: Reticulocyte Count
Description: Reticulocytes are immature red blood cells.
Time Frame: Baseline, Week 1, Week 2, Week 4 and Week 8
Population: Participants who received erythropoietin treatment and had the data available at least on Baseline and at all measurable time points of study evaluation period. Here, 'N' signifies participants who were evaluablated for this outcome measure and 'n' signifies participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 18
Nanogram per liter
  Baseline (n=18) | 92.33 (58.27)
  Week 1 (n=17) | 64.81 (83.90)
  Week 2 (n=16) | 200.74 (110.37)
  Week 4 (n=17) | 120.68 (118.18)
  Week 8 (n=7) | 111.74 (70.37)

7. Secondary Outcome: Serum Ferritin Level
Description: Serum ferritin is the amount of ferritin in a participant's blood. Ferritin is a protein that stores iron and allows the body to use iron.
Time Frame: Baseline, Week 1 and Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Microgram per liter
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 19
Microgram per liter
  Baseline (n=19) | 807.28 (746.84)
  Week 1 (n=18) | 870.28 (638.48)
  Week 2 (n=18) | 685.11 (565.32)

8. Secondary Outcome: Serum Iron Level
Description: Serum iron is a test that measures the amount of iron in the blood which is bound to transferrin.
Time Frame: Baseline, Week 1 and Week 2
Population: Participants who received erythropoietin treatment and had the data available at least on Baseline and at all measurable time points of study evaluation period. Here, 'N' signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Microgram per deciliter (Mcg per dl)
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 18
Microgram per deciliter (Mcg per dl)
  Baseline | 66.06 (65.04)
  Week 1 | 89.22 (74.35)
  Week 2 | 53.06 (31.74)

9. Secondary Outcome: Transferring Iron Binding Capacity (TIBC)
Description: TIBC is a medical laboratory test that measures the blood's capacity to bind iron with transferrin.
Time Frame: Baseline, Week 1 and Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Mcg per dl
Arm/Group | Participants With Cancer Related Anemia
Number analyzed (Participants) | 19
Mcg per dl
  Baseline (n=19) | 275.26 (54.62)
  Week 1 (n=18) | 281.39 (54.75)
  Week 2 (n=18) | 288.17 (65.39)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 8
Description: Participants evaluated for safety included all the participants who received erythropoietin treatment and who had sufficient data to perform statistical evaluation.
Arm/Group | Participants With Cancer Related Anemia
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Cancer Related Anemia (N=25)
Vomitting (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Cancer Related Anemia (N=25)
Leukopenia (Blood and lymphatic system disorders) | 4
Skin rash (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2
Insomnia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Mucosal inflammation (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Fatigue (General disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Blood creatinine increased (Investigations) | 1
Herpes zoster (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Tremor (Nervous system disorders) | 1
Palpitation (Cardiac disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Haemoglobinaemia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No